CLINICAL TRIAL: NCT00141999
Title: An Evaluation of Long-Term Protection Against Hepatitis B Virus Infection: Response of Alaska Native Children and Adolescents Who Received the Primary Recombinant Hepatitis B Vaccine Series Beginning at Birth to an Additional Dose of Vaccine
Brief Title: Response to Booster Doses of Hepatitis B Vaccine in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Alaska Native Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CDC-NCID-2998; U50/CCU022279
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Hepatitis
Keywords: vaccine; hepatitis
MeSH Terms: conditions — Hepatitis | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: hepatitis B vaccine

SUMMARY:
The purpose of this study is to determine the immune response to an additional (booster) dose of hepatitis B vaccine 5-14 years after a three dose series was given

DETAILED DESCRIPTION:
Routine hepatitis B vaccination beginning at birth was provided to Alaska Natives several years before other areas of the United States began routine infant hepatitis B vaccination programs. Follow up studies of hepatitis B immunity among Alaska Native children provide an early opportunity to assess long term protection against hepatitis B virus (HBV) infection for children vaccinated at birth with the currently used recombinant vaccine. This protocol describes an evaluation of long-term protection against HBV infection among children who received the recombinant hepatitis B vaccine beginning at birth, and who currently receive medical care at the Alaska Native Medical Center (ANMC) in Anchorage, Alaska.

The specific objective of this study is to evaluate the immune response to a five microgram dose of recombinant hepatitis B vaccine among 5-6 year old and 10-14 year old children who received the primary recombinant hepatitis B vaccine series beginning at birth. The concentration of antibodies to hepatitis B surface antigen (anti-HBs) will be measured immediately before administering the vaccine, and compared with levels in serum drawn 1, 2 and 4 weeks afterwards. A rapid antibody response (anamnestic response) indicates that immune memory, and therefore immunity to HBV infection, is preserved. The frequency and magnitude of the anamnestic response for the group of older children will be compared to that of the younger group.

Currently, there is no recommendation for a routine booster dose of vaccine after receiving three doses at birth. This study will provide valuable information regarding the need for and response to an additional dose (booster dose) of hepatitis B vaccine among children entering primary school or adolescence. If evidence of waning immune memory (as measured by a delayed or diminished response to the additional dose of vaccine) is found, these two age groups would be the most easily accessible for routine delivery of a booster dose.

ELIGIBILITY:
Inclusion Criteria:

Received 3 doses of hepatitis B vaccine during infancy, beginning at birth

Exclusion Criteria:

Mother HBsAg-positive immunosuppressed

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400
Dates: Start 2001-05; Primary Completion 2005-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Fiore, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Alaska Native Medical Center, Anchorage, Alaska, United States